CLINICAL TRIAL: NCT02128165
Title: Effect of Gastric Balloon in Morbid Obesity: Prospective Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, MOHAMED ABDELLATIF, phd, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Air gastric balloon
Record Dates: First submitted 2014-04-26; First posted 2014-05-01 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Morbid Obesity
Keywords: gastric balloon; morbid obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMI more than 45 BMI (Active Comparator): Air filled gastric balloon (Heliosphere) those BMI above 45
  Interventions: Device: BMI more than 45 BMI
- BMI less than 45 BMI (Active Comparator): Air filled gastric balloon (Heliosphere)those BMI below 45
  Interventions: Device: BMI less than 45 BMI

INTERVENTIONS:
Device: BMI more than 45 BMI — Air filled gastric balloon (Heliosphere) those BMI above 45
  Arms: BMI more than 45 BMI
Device: BMI less than 45 BMI — Air filled gastric balloon (Heliosphere) those BMI below 45
  Arms: BMI less than 45 BMI

SUMMARY:
The aim of this study is to compare the efficacy of gastric balloon in weight reduction among two different categories of morbidly obese people.

DETAILED DESCRIPTION:
To study to effect of gastric balloon in weight reduction among those above 35 BMI and those above 45 BMI.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity

Exclusion Criteria:

* patient refusal
* psychological patients
* oesophageal or gastric abnormalities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Effect of weight loss | 6 months
  By following up the BMI every month

SECONDARY OUTCOMES:
Tolerance | 6 months
  Tolerance of patients to the balloon in form of vomiting, nausea, gastric pain

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt